CLINICAL TRIAL: NCT04781166
Title: An Online Intervention to Reduce Self-Harm Among Persons With High Emotion-Related
Brief Title: An Online Intervention to Reduce Self-Harm Among Persons With High Emotion-Related Impulsivity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Sheri L. Johnson, Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UC CPHS 2016-01-8287
Record Dates: First submitted 2021-02-19; First posted 2021-03-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Suicidal Ideation; Deliberate Self-harm; Impulsivity
MeSH Terms: conditions — Suicidal Ideation; Self-Injurious Behavior; Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: Adult participants will be enrolled in the intervention, and we will use pre-, post-data to evaluate whether the program appears to be helpful. Adolescent participants will be randomly assigned to a waitlist control or intervention; those in the waitlist will be offered the intervention after they complete the waitlist period.
Who Masked: Outcomes Assessor
Masking Description: Interview-based assessments will be conducted by personnel who are unaware of treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be immediately assigned to the intervention.
  Interventions: Behavioral: Calm program
- Waitlist control (Other): Participants will complete measures before and after a waitlist equivalent to the duration of the intervention, to assess whether change is observed with time and repeated assessment. After the waitlist control, participants will be provided the opportunity to take part in the intervention. In this RDICT design, the pre- post- treatment data will be included in analyses.
  Interventions: Behavioral: Calm program

INTERVENTIONS:
Behavioral: Calm program — 7 online modules designed to teach cognitive behavioral skills

SUMMARY:
The goal of this program is to test a brief, online, cognitive behavioral intervention for people who struggle with self-harm or suicidal urges or behavior in the context of emotion-related impulsivity.

DETAILED DESCRIPTION:
Participants will be asked to complete 7 brief online modules to cover how to understand emotion-triggered impulsivity, to better detect states of high emotion and arousal, to learn new strategies for self-calming high arousal, and to pre-plan how to cope with high arousal states. As part of the program, participants receive daily texts and prompts to remind them of the intervention content and skills. At baseline and follow-up, participants will complete measures of emotion-related impulsivity, self-harm, and suicidality.

ELIGIBILITY:
Inclusion Criteria:

* at least 13 years of age
* engaged in mental health care
* evidence of either self-harm or suicidal urges or behavior in the past 3 months
* high levels of emotion-related impulsivity.

Exclusion Criteria:

* inability to adequately take part in the online measures due to problems with intellectual function, language, or other conditions,
* psychosis,
* not currently living in California,
* lack of access to a device to privately complete online modules.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in suicidal ideation among adults | immediately before the intervention and one week after intervention
  Columbia Suicide Severity Rating scale suicidal ideation severity score; scores range from 0 to 5, where 5 is more severe.
Change in interview-rated suicidal ideation among adolescent patients | immediately before the intervention and one week after intervention
  Self-Injurious Thoughts and Behaviors Interview suicidal ideation in the past month scored as the sum of the items on the worst intensity, average intensity, and likelihood of suicidal ideation items; scores range from 0 to 12, with higher scores reflecting greater severity.
Change in self-rated suicidal ideation among adolescent patients | immediately before the intervention and one week after intervention
  Suicide Ideation Questionnaire Jr; scores range from 0 to 6, where 6 is more severe
Change in self-rated deliberate self-harm | immediately before the intervention and one week after intervention
  Deliberate Self-Harm Inventory Frequency in past month score, from 0 to number of incidents reported (higher scores are worse outcomes)
Change in interview-based self-harm among adolescent patients | immediately before the intervention and one week after intervention
  Self-Injurious Thoughts and Behaviors Interview NSSI severity in the past month, scored as the sum of the items on the worst intensity, average intensity, and likelihood of NSSI items; scores range from 0 to 12 with higher scores reflecting greater severity.
Change in impulsivity | immediately before the intervention and one week after intervention
  self-rated Three factor impulsivity Feelings Trigger Action subscale; scores range from 1 to 5, where 5 reflects more severe impulsivity
Change in interview-based impulsivity among adolescent patients | immediately before the intervention and one week after intervention
  Urgency interview scores, scored as the sum of 8 items, range = 0 to 16, where higher scores reflect more impulsivity.

SECONDARY OUTCOMES:
Change in aggression | immediately before the intervention and one week after intervention
  Bryant Aggression scale: mean of physical aggression, verbal aggression, and anger subscales; range of scores from 1 to 5, where 5 = more severe aggression

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L Johnson, Ph.D., Principal Investigator — professor
Locations (1):
- University of California, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide fully de-identified data on OSF.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will upload data at the time we submit the article for publication. Data will be available for 7 years.
Access Criteria: Data will be available to authorized users of the OSF website.